CLINICAL TRIAL: NCT04195113
Title: Management and Outcomes of Patients Receiving Oral Anticoagulants Who Require an Urgent/Emergency Surgery or Procedure: A Prospective Registry Study
Brief Title: Perioperative Anticoagulant Use for Surgery Evaluation Emergency Registry
Acronym: PAUSE-ER
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Deborah Siegal, Dr. Deborah Siegal - Principal Investigator, McMaster University
Other Study IDs: PAUSE-ER-2019
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism; Arterial Vascular Disease
Keywords: anticoagulant; atrial fibrillation; venous thromboembolism; arterial vascular disease; surgery; oral anticoagulant; blood thinner; warfarin; DOAC; interruption; discontinue; emergency; perioperative; vitamin k antagonist
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Direct Oral Anticoagulants (DOACs): In this study, DOACs include apixaban, dabigatran, edoxaban and/or rivaroxaban.
- Vitamin K Antagonist (VKA): In this study, the VKA is warfarin.

SUMMARY:
Among patients who are receiving long-term anticoagulant therapy, whether with a direct oral anticoagulant (DOAC) or vitamin K antagonist (VKA), approximately 3-5% who require treatment interruption for a surgery will do so in an urgent/emergency surgery setting. Additionally, there is considerable morbidity and mortality associated with DOAC/VKA management in an urgent/emergency surgery setting. Thus, this prospective registry study aims to identify and compare determinants for perioperative adverse events in DOAC-treated and VKA-treated patients who require an urgent/emergency surgery, and to identify which of these are modifiable. It also aims to describe and compare management of anticoagulant reversal (i.e., non-specific and specific reversal agents) and resource utilization (i.e., blood transfusion) in DOAC- and VKA-treated patients who need an urgent/emergency surgery.

DETAILED DESCRIPTION:
Among patients who are receiving long-term anticoagulant therapy, whether with a direct oral anticoagulant (DOAC) or vitamin K antagonist (VKA), approximately 3-5% who require treatment interruption for a surgery will do so in an urgent/emergency surgery setting. Assuming that approximately 500,000 to 800,000 patients per year in the U.S. and E.U. will require perioperative management for a surgery/procedure, the investigators estimate that approximately 20,000 to 25,000 patients will require an urgent/emergency surgery. Although this represents a small proportion of patients who require anticoagulant interruption, there is considerable morbidity and mortality associated with DOAC/VKA management in an urgent/emergency surgery setting. Thus, for VKA-treated patients, rates of thromboembolism, major bleeding and mortality are 10.5%, 22.9%, and 2.9%, respectively. Similarly, for DOAC-treated patients who require an urgent/emergency surgery, rates of thromboembolism, major bleeding and mortality are 7.4%, 17.6%, and 1.5%, respectively. By comparison, rates of these outcomes for DOAC/VKA-treated patients who need elective surgery are ~0.5-1.0%, ~1-3%, and <0.5%, respectively. Most studies have focused on the perioperative anticoagulant management of patients who require an elective surgery/procedure. To the investigators' knowledge, few studies have focused on the assessment of adverse outcomes in an urgent/emergency perioperative setting among anticoagulated patients. Thus, this prospective registry study aims to 1) identify and compare determinants for perioperative adverse events in DOAC-treated and VKA-treated patients who require an urgent/emergency surgery, and to identify which of these are modifiable, and 2) describe and compare management of anticoagulant reversal (i.e., non-specific and specific reversal agents) and resource utilization (i.e., blood transfusion) in DOAC- and VKA-treated patients who need an urgent/emergency surgery. The data gained from this study will generate hypotheses for subsequent prospective studies that would potentially assess different management strategies in this clinical setting (e.g., use of DOAC antidote- vs. prothrombin complex concentrate-based management).

Given the exploratory, hypothesis-generating nature of the proposed study, the sample size is one of convenience, comprising 200 DOAC- and 200 warfarin-treated patients. Patients will be recruited from 30 clinical sites in Canada, the US, and Europe. With 30 clinical sites, the investigators estimate that 3-5 patients/month (60-72/yr) per arm can be recruited, corresponding to an overall rate of 180-216 over 3 years. Each study patient will participate for approximately 4 weeks, with one follow-up phone call at 4 weeks post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years) receiving a DOAC (dabigatran, rivaroxaban, apixaban or edoxaban) or a VKA (warfarin) for stroke prevention atrial fibrillation/flutter, treatment or secondary prevention of venous thromboembolism or treatment of arterial vascular disease.
* Requires an urgent or emergency surgery and planned surgery is scheduled within 72 hours from the time the decision was made to proceed to surgery (e.g. time of assessment in emergency department, or time of consultation note etc.) or if the time of the decision to proceed to surgery is unavailable, from the time from admission to surgery; or urgent surgery as deemed by Investigator.
* Patient or delegate is willing and able to provide written informed consent while patient is hospitalized and agree to telephone follow-up 30 days (±7 days) after surgery.

Exclusion Criteria:

* Patient receiving a non-warfarin VKA.
* Patient enrolled in the study previously and had the urgent procedure/surgery (if procedure/surgery cancelled, patient can re-enroll)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study cohort will be recruited from urgent care and/or emergency department populations.
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who had arterial thromboembolism (ATE) | Each patient will be followed-up once 30±7-days post-operative
  Any of the following: stroke, systemic arterial embolism, and/or myocardial infarction.
  * Ischemic stroke: any new focal neurologic deficit that persists for >24 hours or any new focal neurologic deficit of any duration, that occurs with evidence of acute infarction on computed tomography (CT) or magnetic resonance imaging (MRI) of the brain.
  * Systemic embolism: symptomatic embolism to upper or lower extremity or abdominal organ, confirmed intraoperatively or by objective imaging (e.g., CT angiography).
  * Myocardial Infarction: Symptomatic myocardial ischemia, defined by pre-specified clinical and objective EKG- and/or troponin-related criteria.
Number of patients who had venous thromboembolism (VTE) | Each patient will be followed-up once 30±7-days post-operative
  Any of the following: symptomatic deep vein thrombosis and/or pulmonary embolism, confirmed by objective imaging studies (e.g., ultrasound, CT pulmonary angiogram, VQ scan).
Number of patients who had major bleeding | Each patient will be followed-up once 30±7-days post-operative
  As defined by the International Society on Thrombosis and Haemostasis (ISTH), ≥1 of the criteria below:
  * bleeding that is fatal or is symptomatic and retroperitoneal, intracranial, intraspinal, intraocular, pericardial, intramuscular with compartment syndrome, or intra-articular
  * non-surgical bleeding causing a drop in hemoglobin ≥20 g/L (1.24 mmol/L) or leading to transfusion ≥2 units whole blood or red cells within 48 hours of the bleed
  * surgical bleed that leads to intervention (e.g., re-operation) or has one of: (i) interferes with mobilization; (ii) leads to delayed wound healing; or (iii) leads to deep wound infection
  * surgical site bleeding that is unexpected and prolonged and/or sufficiently large to cause hemodynamic instability associated with: (i) drop in hemoglobin ≥20 g/L (1.24 mmol/L); or (ii) transfusion of ≥2 units whole blood or red cells within 48 hours of the bleed
Number of patients who died | Each patient will be followed-up once 30±7-days post-operative
  Death due to any cause

SECONDARY OUTCOMES:
Number of patients who received adjunctive hemostatic therapies | Each patient will be followed-up once 30±7-days post-operative
  For example, prothrombin complex concentrates, FEIBA, tranexamic acid, etc.
Number of patients who received specific anticoagulant reversal agents | Each patient will be followed-up once 30±7-days post-operative
  For example, idarucizumab (for dabigatran), andexanet alfa (for factor Xa inhibitors), vitamin K (for VKA), prothrombin complex concentrates (for VKA) etc.
Number of patients who received blood products | Each patient will be followed-up once 30±7-days post-operative
  For example, packed red blood cells, platelets, plasma, cryoprecipitate, fibrinogen, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Siegal, MD MSc FRCPC, Principal Investigator — McMaster University; James Douketis, MD MSc FRCPC, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario